CLINICAL TRIAL: NCT07085338
Title: A Phase II Study With a Safety Run-In of the Addition of N-803, a Novel IL-15 Super-Agonist, to a Chemoimmunotherapy Backbone for the Treatment of Patients With Relapsed or Refractory Neuroblastoma
Brief Title: A Phase II Study With a Safety Run-In of the Addition of N-803 to a Chemoimmunotherapy Backbone for the Treatment of Patients With Relapsed or Refractory Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HuNB803; NCI-2025-02707 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2025-04-09; First posted 2025-07-25 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Neuroblastoma Recurrent
Keywords: relapse; refractory
MeSH Terms: conditions — Recurrence | interventions — Temozolomide; Irinotecan; Hu14.18K322A monoclonal antibody; ALT-803; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Chemoimmunotherapy (Experimental): Patients will be randomized to receive chemoimmunotherapy alone.
  Interventions: Drug: Temozolomide; Drug: Irinotecan; Drug: hu14.18K322A; Drug: Sargramostim
- Chemoimmunotherapy + N-803 (Experimental): Patients will be randomized to receive chemoimmunotherapy plus N-803.
  Interventions: Drug: Temozolomide; Drug: Irinotecan; Drug: hu14.18K322A; Drug: N803; Drug: Sargramostim
- Safety Run-In Treatment Schedule - Chemoimmunotherapy + N-803 (Experimental): The first 6 patients included in the safety assessment run-in phase will receive cycles of irinotecan, temozolomide, hu14.18K322A, GM-CSF and N-803. If fewer than 2 patients in the first cohort of 6 patients experience a DLT in Cycle 1, then the trial will proceed to Phase 2. If 2 or more of the first 6 patients experience a DLT in Cycle 1 then the N-803 will be dose reduced to 15 mcg/kg and 6 more patients will be enrolled in the safety assessment run-in.
  Once the safety assessment run-in phase is completed, patients will be enrolled onto the phase 2 study.
  Interventions: Drug: Temozolomide; Drug: Irinotecan; Drug: hu14.18K322A; Drug: N803; Drug: Sargramostim

INTERVENTIONS:
Drug: Temozolomide — IV, Days 1-5
Drug: Irinotecan — IV, Days 1-5
Drug: hu14.18K322A — IV over 4 hours daily times 4 doses, Days 2-5.
Drug: N803 — Subcutaneous (SC), Day 6.
  Arms: Chemoimmunotherapy + N-803; Safety Run-In Treatment Schedule - Chemoimmunotherapy + N-803
Drug: Sargramostim — Subcutaneous injection (preferred) or IV, Days 7-13.
  Other Names: GMCSF

SUMMARY:
The study participant is being asked to take part in this research study because the participant has been diagnosed with neuroblastoma that did not fully respond to previous treatment (refractory), or it has returned after treatment (relapsed).

Primary Aims

* To evaluate if the administration of N-803 in combination with irinotecan, temozolomide, hu14-18K322A, and GM-CSF in patients with relapsed/refractory neuroblastoma is feasible and tolerable
* To determine if the response rate of N-803 with irinotecan, temozolomide, hu14.18K322A and GM-CSF in patients with relapsed/refractory neuroblastoma is superior to the combination of irinotecan, temozolomide, hu14.18K322A, and GM-CSF

Secondary Aims

* To describe the toxicity profile of N-803 administered with irinotecan, temozolomide, hu14.18K322A and GM-CSF
* To evaluate and compare the progression free survival (PFS) and overall survival (OS) of and between patients receiving irinotecan, temozolomide, hu14.18K322A and GM-CSF with and without N-803

DETAILED DESCRIPTION:
This is a randomized phase 2 study with a safety assessment run-in conducted in children with relapsed or refractory neuroblastoma to evaluate the feasibility, tolerability, and response to chemoimmunotherapy backbone (irinotecan, temozolomide, hu14.18K322A and GM-CSF) with or without N-803. The first 6 patients included in the safety assessment run-in phase will receive irinotecan, temozolomide, hu14.18K322A, GM-CSF and N-803. If fewer than 2 patients in the first cohort of 6 patients experience a DLT in Cycle 1, then the trial will proceed Phase 2. If 2 or more of the first 6 patients experience a DLT in Cycle 1 then the N-803 will be dose reduced, and 6 more patients will be enrolled in the safety assessment run-in.

Once the safety assessment run-in phase is completed, patients will be enrolled onto the phase 2 study. In the phase 2 study, patients will be randomized to receive either chemoimmunotherapy alone (Arm A) or chemoimmunotherapy plus N-803 (Arm B). Patients treated on Arm A who experience disease progression may cross over at any time point after completing Cycle 2 and receive therapy administered on Arm B. Pharmacokinetic and correlative biology studies will be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Age

- Patients must be < 30 at the time of enrollment on study.

Diagnosis

- Patients must have had histologic verification of neuroblastoma or demonstration of neuroblastoma cells in the bone marrow with elevated urinary or serum catecholamines [i.e., > 2 x upper limit of normal (ULN)], at the time of initial diagnosis.

Disease Risk Group

* Patients must have high-risk neuroblastoma according to COG risk classification at the time of study registration. Patients whose disease was initially considered low or intermediate risk but were then reclassified as high-risk neuroblastoma prior to enrollment are also eligible.

Response to Prior Therapy (using INRC definitions)

- Patients must have at least ONE (recurrent/progressive, refractory, or persistent) of the following:

* Recurrent/progressive disease after the diagnosis of high-risk neuroblastoma at any time prior to enrollment regardless of response to frontline therapy. (Note that this excludes patients initially considered low or intermediate risk that progressed to high-risk disease but have not progressed after the diagnosis of high-risk neuroblastoma).
* Refractory disease: A best overall response of no response/stable disease since diagnosis of high-risk neuroblastoma AND after at least 4 cycles of induction therapy.
* Persistent disease: A best overall response of partial response since diagnosis of high-risk neuroblastoma AND after at least 4 cycles of induction therapy

Sites of Disease

- Patients must have at least ONE of the following (lesions may have received prior radiation therapy if they meet the other criteria listed below) based on institutional assessment:

Bone Sites

• MIBG avid tumors: patients must meet one of the following criteria:

a. Patients with recurrent/progressive or refractory disease: i. Must have at least one MIBG avid bone site on planar imaging OR ii. Must have > 2 lesions on SPECT/CT. A biopsy is not required unless the above imaging criteria are not met

b. Patients with persistent disease: i. If a patient has 3 or more MIBG avid bone lesions, then no biopsy is required.

ii. If a patient has only 1 or 2 MIBG avid bone lesion sites, then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one MIBG avid site present at the time of enrollment is required. Bone lesions may be biopsied at any time point prior to enrollment.

* For MIBG non-avid tumors, patients must have at least an FDG-PET avid site and meet the following criteria:

  1. Biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma at any time prior to enrollment of at least one FDG-PET avid site.

     Bone Marrow

     - Any amount of tumor cells in the bone marrow (including neuroblasts, mature and maturing ganglion cells) done at the time of study enrollment based on routine morphology and/or immunohistochemistry in at least one sample from bilateral aspirates and biopsies. NOTE: Patients with bone marrow disease only will be eligible if they have more than 5% disease involvement (documented neuroblastoma cells) in at least one sample from bilateral bone marrow biopsies.

     Soft Tissue Sites

     - At least one soft tissue lesion that meets criteria for a TARGET lesion as defined by:
* SIZE: Lesion can be accurately measured in at least one dimension with a longest diameter ≥ 10 mm, or for discrete lymph nodes ≥ 15mm on short axis. Lesions meeting size criteria will be considered measurable.
* In addition to size, a lesion needs to meet ONE of the following criteria except for patients with parenchymal CNS lesions which will only need to meet size criteria:

  a. For MIBG avid tumors: lesion must be MIBG avid and meet one of the following criteria: i. For patients with recurrent/progressive or refractory disease: no biopsy is required ii. For patients with persistent disease:
* If a patient has 3 or more MIBG avid soft tissue lesions, then no biopsy is required.
* If a patient has only 1 or 2 MIBG avid soft tissue lesion sites) then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one MIBG avid site present at the time of enrollment is required. Soft tissue lesions may be biopsied at any time point prior to enrollment.

  b. For MIBG non-avid tumors patient must have at least one FDG avid site and meet the following criteria: i. Biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma from a lesion at any time prior to enrollment of at least one FDG-PET avid site.

ii. At least one non-target soft tissue lesion that is not measurable but had a biopsy positive for neuroblastoma and/or ganglioneuroblastoma at any time prior to enrollment OR is MIBG avid on planar imaging.

Patients with elevated catecholamines (i.e., > 2 x ULN) only are NOT eligible for this study.

Performance Status

- Patients must have Lansky (≤16 years) or Karnofsky (>16 years) score of ≥50 (Appendix I).

Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Prior Therapy

- Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study registration. Patients must not have received the therapies indicated below within the specified time prior to registration on this study as follows:

Table 2: Prior Therapies List Type of Therapy Specified Time Period Additional Comments Myelosuppressive Chemotherapy ≤ 14 days This includes cytotoxic agents given on a low dose metronomic regimen as well as retinoids.

Biologic Antineoplastic (anti-neoplastic agents)1 ≤ 7 days Monoclonal Antibodies ≤ 7 days or 3 half-lives whichever is longer, but no longer than 30 days (with recovery of any associated toxicities).

Cellular Therapy (e.g., modified T cells, NK cells, dendritic cells, etc.) ≤ 21 days and with recovery of all associated toxicities Radiation Small port radiation ≤ 7 days Large field radiation therapy ≤ 12 weeks i.e., total body irradiation, craniospinal, whole abdominal, total lung, > 50% marrow space Other Substantial Bone Marrow Radiation ≤ 6 weeks 131I-MIBG therapy ≤ 6 weeks Hematopoietic Stem Cell Transplant Autologous Stem Cell Infusion Following Myeloablative Therapy ≤ 6 weeks Patients who have received an autologous stem cell infusion to support non-myeloablative therapy (such as 131I-MIBG) are eligible at any time as long as they meet the other criteria for eligibility.

Any other investigational agents (covered under another IND) ≤ 14 days

1. Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or ANC counts)

   Concomitant Therapy Restrictions
   * Patients must not have received the concomitant medications indicated below within the specified time prior to study registration or planned treatment start date on this study as follows:

     • No other anti-cancer agents or radiotherapy at the time of study registration or while on study.

     • No short-acting hematopoietic growth factors within 7 days of blood draw documenting eligibility and no long-acting hematopoietic growth factors within 14 days of blood draw documenting eligibility.

     • Patients must not have received 0.5 mg/kg/day (prednisone equivalent) doses of systemic steroids for at least 7 days prior to study enrollment.

     • Inhaled steroids are permitted to treat reactive airways

     • < 2mg/kg of hydrocortisone or equivalent is permitted as blood product premedication to avoid allergic reactions.

     • Physiologic hydrocortisone dosing is permitted for patients with known adrenal insufficiency.

     • The use of dexamethasone as an antiemetic is not permitted.
     * Irinotecan is a substrate for CYP3A4 (major) and CYP2B6 (major). Patients who have received drugs that are strong inducers or inhibitors of CYP3A4 within 7 days prior to study enrollment are not eligible. The use of strong inducers or inhibitors of CYP3A4 (Appendix II) and CYP2B6 (e.g., carbamazepine) should be avoided for the duration of protocol therapy. Consult drug information references for further information. In addition, concomitant use of BCRP inhibitors (cyclosporine, eltrombopag, gefitinib), and UGT1A1 inhibitors (diclofenac, ketoconazole, probenecid, silibinin, nilotinib, and atazanavir) should be avoided due to potential increased risk of irinotecan toxicity.

       * Moderate inducers or inhibitors of CYP3A4 (Appendix II) should also be avoided during protocol therapy if reasonable alternatives exist.

   Organ Function Requirements

   Hematologic Function:
   * Patients must meet the following hematologic criteria for enrollment regardless of bone marrow disease involvement:

     1. ANC ≥750/μL, (no short-acting hematopoietic growth factors ≤ 7 days of blood draw documenting eligibility and no long-acting hematopoietic growth factors ≤ 14 days of blood draw documenting eligibility); and
     2. Platelet count ≥ 75,000/μL, transfusion independent (no platelet transfusions ≤ 7 days of blood draw documenting eligibility).

   Renal Function

   a. Patients must have adequate renal function defined as age-adjusted serum creatinine ≤1.5 ULN for age (see below):

   Table 3: Age-Adjusted Serum Creatinine Age Maximum Serum Creatine (mg/dL) Male Female

1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4 > 16 years 1.7 1.4

Liver Function

1. Total bilirubin ≤ 1.5 x ULN for age; and,
2. SGPT (ALT) ≤ 225 U/L (≤ 5x ULN). Note that for ALT, the upper limit of normal for all sites is defined as 45 U/L.

Cardiac Function

1. Shortening fraction of ≥ 27% by ECHO, or
2. Ejection fraction of ≥ 50% by ECHO or gated radionuclide study.

Pulmonary Function

No evidence of dyspnea at rest, no exercise intolerance.

Adequate Central Nervous System Function

1. Patients with a history of CNS disease must have no clinical or radiological evidence of active CNS disease at the time of study enrollment
2. Patients with seizure disorders may be enrolled if seizures are well controlled on anti-seizure medications
3. CNS toxicity ≤ Grade 2

   Reproductive Function
   * All post-menarchal females must have a negative serum or urine beta-HCG ≤ 7 days prior to registration. Male and female subjects of reproductive age and childbearing potential must agree to use two acceptable methods of birth control (i.e., intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) or to abstain from heterosexual intercourse for the duration of their participation in the study.

   Central Nervous System (CNS)

   - Patients with a history of intraparenchymal or leptomeningeal based CNS disease must have no clinical or radiological evidence of active CNS disease at the time of study enrollment.

   - Patients with skull-based tumors with direct intracranial extension are eligible if there are no neurologic signs or symptoms related to the lesion.

   Exclusion Criteria:

   - Pregnancy, breast feeding, or unwillingness to use effective contraception during the study will not be entered on this study due to risks of fetal and teratogenic adverse events. Females of childbearing potential must have a negative pregnancy test to be eligible for this study.

   - Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

   - Patients with disease of any major organ system that would compromise their ability to withstand therapy.

   - Patients who have undergone a prior allogeneic stem cell or solid organ transplant.

   - Patients who are on hemodialysis.

   - Patients with an active or uncontrolled infection. Patients on prolonged antifungal therapy are still eligible if they are culture negative, afebrile, and meet other organ function criteria.

   - Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C. Testing is not required in the absence of clinical findings or suspicions.

   - Patients who require or are likely to require pharmacologic doses of systemic corticosteroids while receiving treatment on this study are ineligible. The only exception is for patients known to require 2 mg/kg or less of hydrocortisone (or an equivalent dose of an alternative corticosteroid) as premedication for blood product administration in order to avoid allergic transfusion reactions. The use of conventional doses of inhaled steroids for the treatment of reactive airway disease is permitted, as is the use of physiological doses of steroids for patients with known adrenal insufficiency.

   - Patients on any other immunosuppressive medications (e.g., cyclosporine, tacrolimus) are not eligible.

   - Patients must not have received enzyme-inducing anticonvulsants including phenytoin, phenobarbital, or carbamazepine for at least 7 days prior to study enrollment. Patients receiving non-enzyme inducing anticonvulsants such as gabapentin, valproic acid, or levetiracetam will be eligible.

   - Patients who have received drugs that are strong inducers or inhibitors of CYP3A4 within 7 days prior to study enrollment are not eligible.

   - Patients must not have been diagnosed with myelodysplastic syndrome or with any malignancy other than neuroblastoma.

   - Patients with symptoms of congestive heart failure are not eligible.

   - Patients must not have > Grade 2 diarrhea.
   * Patients with a history of progressive disease while receiving therapy per ANBL1221.
   * Patients with a history of Grade 4 allergic reactions to anti-GD2 antibodies or reactions that required permanent discontinuation of the anti-GD2 therapy are not eligible.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate if the administration of N-803 in combination with irinotecan, temozolomide, hu14-18K322A, and GM-CSF in patients with relapsed/refractory neuroblastoma is feasible | Complete Cycle 1 treatment (each cycle is 21 days)
  Feasibility Measures: Patients evaluable for toxicity in the safety run-in must receive one dose of N-803. The proportion of evaluable patients who successfully complete the protocol-defined treatment regimen in the Safety Run-in phase will be calculated. The reasons for treatment discontinuation or deviations from the protocol will be summarized.
To determine if the response rate of N-803 with irinotecan, temozolomide, hu14.18K322A and GM-CSF in patients with relapsed/refractory neuroblastoma is superior to the combination of irinotecan, temozolomide, hu14.18K322A, and GM-CSF | Complete Cycle 1 treatment (each cycle is 21 days)
  Tolerability Assessments: Tolerability of the protocol-defined treatment in the Safety Run-in phase will be determined by assessing adverse events and their severity. Adverse events will be categorized based on standard CTCAE v5.0 criteria. Dose modifications or interruptions resulting from treatment-related adverse events will be analyzed.
To determine if the response rate of N-803 with irinotecan, temozolomide, hu14.18K322A and GM-CSF in patients with relapsed/refractory neuroblastoma is superior to the combination of irinotecan, temozolomide, hu14.18K322A, and GM-CSF | Up to 10 cycles of irinotecan/temozolomide/hu14.18K322A/GM-CSF with or without N-803 in the Phase 2 (each cycle is 21 days)
  Tumor response will be assessed using standard NANT criteria. The primary endpoint for response analysis will be Best Overall Response (BOR), defined as the best response observed prior to progression, cross over or start of another therapy. Point estimates for the response rate (proportion of patients who have BOR of PR or better) will be calculated, together with exact 95% confidence intervals.

SECONDARY OUTCOMES:
To describe the toxicity profile of N-803 administered with irinotecan, temozolomide, hu14.18K322A and GM-CSF | Up to 10 cycles of irinotecan/temozolomide/hu14.18K322A/GM-CSF with or without N-803 in the Phase 2 (each cycle is 21 days)
  Toxicities will be graded using CTCAE v5.0. The toxicity profile will be defined as a comprehensive assessment of adverse events, categorized by standard toxicity criteria. The frequency, type, and severity and attribution of adverse events will be calculated and summary statistics for the toxicity profile will be provided.
To evaluate and compare the progression free survival (PFS) of and between patients receiving irinotecan, temozolomide, hu14.18K322A and GM-CSF with and without N-803 | Time from enrollment (phase I) or randomization (phase II) to disease progression, death, or last follow-up, whichever is earlier, assessed up to 36 months
  Progression-Free Survival (PFS) is defined as the time from the start of treatment to disease progression or death from any cause. Time from the day of receiving irinotecan, temozolomide, hu14.18K322A and GM-CSF with and without N-803 to the day of development of any progression or death will be assessed by the Kaplan-Meier method separately. The PFS rate will be estimated along with the corresponding 95% CI. A log-rank test will be used to compare between the two groups with and without N-803.
To evaluate and compare overall survival (OS) of and between patients receiving irinotecan, temozolomide, hu14.18K322A and GM-CSF with and without N-803 | Time from date of enrollment (phase I) or randomization (phase II) until the date of death from any cause, or last follow-up, whichever is earlier, assessed up to 36 months.]
  Overall Survival (OS) is defined as the time from the start of treatment to death from any cause. Time from the day of receiving irinotecan, temozolomide, hu14.18K322A and GM-CSF with and without N-803 to the day of development of any progression or death will be assessed by the Kaplan-Meier method separately. The OS rate will be estimated along with the corresponding 95% CI. A log-rank test will be used to compare between the two groups with and without N-803.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Federico, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols